CLINICAL TRIAL: NCT06632080
Title: Effects of Substance P on Headache Induction in Healthy Individuals: a Randomized Clinical Trial
Brief Title: Effects of Substance P on Headache Induction in Healthy Individuals
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Håkan Ashina, Senior Researcher, Danish Headache Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: H-23030963
Record Dates: First submitted 2024-10-06; First posted 2024-10-08 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Healthy Volunteers Only
Keywords: Headache
MeSH Terms: conditions — Headache | interventions — Substance P

STUDY DESIGN:
Intervention Model Description: The present trial has a randomized, double-blind, placebo-controlled, 2-way crossover design and will be conducted at a single site.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Substance P (Experimental): Substance P will be administered by intravenous infusion.
  Interventions: Drug: Substance P
- Placebo (Placebo Comparator): Placebo (isotonic saline) will be administered by intravenous infusion.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Substance P — The participants will receive a continuous intravenous infusion of 20 mL of substance P (1.5 pmol/kg/min) over 20 minutes.
  Arms: Substance P
Drug: Placebo — The participants will receive a continuous intravenous infusion of 20 mL of placebo (isotonic saline) over 20 minutes.
  Arms: Placebo

SUMMARY:
Substance P is a signaling molecule that has been implicated in the pathogenesis of headache. This study aims to ascertain whether administration of substance P can induce headache in healthy adults.

DETAILED DESCRIPTION:
Substance P is a vasoactive signaling molecule that belongs to the tachykinin family of peptides. It is expressed in multiple cells, including primary afferents of the trigeminal ganglion that innervate the meninges and its arteries. The best-known function of substance P is its role in pain transmission, and several lines of evidence has implicated substance P in the pathogenesis of headache. This study aims to ascertain whether intravenous infusion of substance P induces headache in healthy individuals who have no past or current history of primary or secondary headache disorder, except for infrequent episodic tension-type headache. For this purpose, we will conduct a randomized, double-blind, placebo-controlled, 2-way crossover trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years of age upon entry into screening
* A body weight of 50 to 100 kg
* Provision of informed consent prior to initiation of any study-specific activities/procedures.

Exclusion Criteria:

* Any history of a primary or secondary headache disorder, except for infrequent episodic tensiontype headache
* Any first-degree relatives with a history of a primary headache disorder, except for infrequent episodic tension-type headache
* Any history of moderate to severe traumatic brain injury
* Any history of cardiovascular disease, including cerebrovascular diseases
* Any history of pulmonary disease
* Any other clinically significant disorders, conditions, or diseases that might impact the safety of the subject or interfere with the study's evaluation, procedures, or completion, aside from those mentioned above. This includes any relevant medical history or evidence that, in the opinion of the site investigator, might pose a risk to the subject or impact the validity of the study results
* The subject is at risk of self-harm or harm to others as evidenced by past suicidal behavior
* Female subjects of childbearing potential with a positive pregnancy test during any study visit
* Cardiovascular disease of any kind, including cerebrovascular diseases
* Hypertension (systolic blood pressure of ≥150 mmHg and/or diastolic blood pressure of ≥100 mmHg) prior to the start of infusion on the experimental day
* Hypotension (systolic blood pressure of ≤90 mmHg and/or diastolic blood pressure of ≤50 mmHg)
* Abnormalities on the electrocardiogram that, in the opinion of the site investigator, might pose a risk to the subject or impact the validity of the study results
* Daily use of any medication other than contraceptives
* Intake of any medication other than contraceptives within 48 hours of infusion start
* Intake of caffeine, nicotine, and alcohol within 12 hours of infusion start
* Headache of any intensity within 48 hours of infusion start

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2024-10-14 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Headache | 12 hours
  The primary outcome is the difference in the incidence of headache* between substance P and placebo during the 12-hour observational period after infusion start.
  * The intensity of headache is rated by the subject on the 11-point numerical rating scale (0 being no headache, 10 being the worst imaginable headache).

SECONDARY OUTCOMES:
Headache Intensity Scores | 12 hours
  The secondary outcome is the difference in the area under the curve for median headache intensity scores between substance P and placebo during the 12-hour observational period after infusion start.

OTHER OUTCOMES:
Dilation of the Superficial Temporal Artery | 2 hours
  The difference in area under the curve for relative STA dilation between substance P and placebo from the start of infusion to 2 hours after the infusion.
Blood Flow Velocity in the Middle Cerebral Artery | 2 hours
  The difference in area under the curve for change in MCA mean blood flow velocity between substance P and placebo from the start of infusion to 2 hours after the infusion.

CONTACTS AND LOCATIONS:
Locations (1):
- Danish Headache Center, Copenhagen University Hospital - Rigshospitalet, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data not published within this article will be made available on reasonable request from any qualified investigator.

REFERENCES:
- [Derived] Al-Khazali HM, Christensen RH, Gozalov E, Hakimzadeh Z, Melchior AG, Dominguez-Moreno R, Ashina M, Ashina H. Effects of substance P on headache induction and arterial dilation in healthy adults. Cephalalgia. 2025 May;45(5):3331024251336132. doi: 10.1177/03331024251336132. Epub 2025 May 14. PMID 40369974